CLINICAL TRIAL: NCT01516892
Title: A Long-term Efficacy, Safety, and Tolerability Study of BOTOX® in Patients With Chronic Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMA-BTX-CM-10-001; The COMPEL Study (Other: Allergan, Inc)
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BOTOX® (Experimental): Participants received 155 U of onabotulinumtoxinA (BOTOX®) approximately every 12 weeks for 108 weeks. OnabotulinumtoxinA was administered as 31 intramuscular injections in 7 head/neck muscle areas.
  Interventions: Biological: onabotulinumtoxinA

INTERVENTIONS:
Biological: onabotulinumtoxinA — Participants received 155 U of onabotulinumtoxinA approximately every 12 weeks for 108 weeks. OnabotulinumtoxinA was administered as 31 intramuscular injections in 7 head/neck muscle areas.
  Other Names: BOTOX®; botulinum toxin Type A

SUMMARY:
This open-label study will assess the long-term efficacy, safety, and tolerability of onabotulinumtoxinA administered for prophylaxis of headaches in patients with chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic migraine (≥15 days per month with headache lasting 4 hours a day or longer)

Exclusion Criteria:

* Diagnosis of myasthenia gravis, Eaton-Lambert Syndrome, or amyotrophic lateral sclerosis
* Headache attributed to another disorder
* Infection or skin disorder at injection sites
* Previous treatment with botulinum toxin of any serotype for any reason
* Anticipated need for botulinum toxin of any type for any reason during the course of the study
* Previous participation in any botulinum toxin clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Actual)
Dates: Start 2011-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (32):
- United States (21):
  - Arizona Neurological Institute, Scottsdale, Arizona
  - The Research Center of Southern California, LLC, Encinitas, California
  - USC Neurology, Los Angeles, California
  - UCSF Headache Center, San Francisco, California
  - Neurological Research Institute, Santa Monica, California
  - Advanced Neurosciences Research, LLC, Fort Collins, Colorado
  - Tampa General Hospital, Tampa, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Robbins Headache Clinic, Northbrook, Illinois
  - Mid-Atlantic Headache Institute, Baltimore, Maryland
  - Kaiser Permanente Research Office/Neurology Department, Largo, Maryland
  - Clinvest Research, Springfield, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Renown Institute for Neurosciences, Reno, Nevada
  - Dent Neurologic Institute, Amherst, New York
  - Montefiore Medical Center, The Bronx, New York
  - Headache Wellness Center, Greensboro, North Carolina
  - Ohio Clinical Research Partners, LLC, Canton, Ohio
  - Jefferson University Hospitals, Philadelphia, Pennsylvania
  - Wesley Headache Clinic, Cordova, Tennessee
  - Baylor Research Institute, Dallas, Texas
- Australia (5):
  - Dr. Joseph Frasca, Adelaide
  - Dr. Con Yiannikas, Burwood
  - Associate Professor Richard Stark, Melbourne
  - Richmmond Neurology, Richmond
  - Associate Professor John O'Sullivan, Spring Hill
- South Korea (6):
  - Hallym University Sacred Heart Hospital, Dongan-gu, Anyang, Anyang Gyeonggi-do
  - Uijeongbu St. Mary's Hospital, Uijeongbu-si, Gyeonggi-do
  - Kangbuk Samsung Hospital, Jongno-Gu, Seoul
  - Seoul St. Mary's Hospital, Jongno-Gu, Seoul
  - Seoul Eulji Hospital, Nowon-Gu, Seoul
  - Yonsei University Dental Hospital, Seodaemum-Gu, Seoul

REFERENCES:
- [Derived] Blumenfeld AM, Charleston L 4th, Kuruvilla D, Savage-Edwards B, Lipton RB, Singh R, Jacob P, Lawrence NA, Wang C, O'Brien HL. OnabotulinumtoxinA treatment among diverse racial groups: Post hoc analysis of the phase 4 Chronic migraine OnabotulinuMtoxinA Prolonged Efficacy open-Label (COMPEL) trial. Headache. 2025 Dec 15. doi: 10.1111/head.70007. Online ahead of print. PMID 41393002
- [Derived] Blumenfeld AM, Tepper SJ, Robbins LD, Manack Adams A, Buse DC, Orejudos A, D Silberstein S. Effects of onabotulinumtoxinA treatment for chronic migraine on common comorbidities including depression and anxiety. J Neurol Neurosurg Psychiatry. 2019 Mar;90(3):353-360. doi: 10.1136/jnnp-2018-319290. Epub 2019 Jan 10. PMID 30630956
- [Derived] Blumenfeld AM, Stark RJ, Freeman MC, Orejudos A, Manack Adams A. Long-term study of the efficacy and safety of OnabotulinumtoxinA for the prevention of chronic migraine: COMPEL study. J Headache Pain. 2018 Feb 5;19(1):13. doi: 10.1186/s10194-018-0840-8. PMID 29404713
- [Derived] Blumenfeld AM, Aurora SK, Laranjo K, Papapetropoulos S. Unmet clinical needs in chronic migraine: Rationale for study and design of COMPEL, an open-label, multicenter study of the long-term efficacy, safety, and tolerability of onabotulinumtoxinA for headache prophylaxis in adults with chronic migraine. BMC Neurol. 2015 Jul 3;15:100. doi: 10.1186/s12883-015-0353-x. PMID 26133547

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BOTOX®
Started | 716
Completed | 373
Not Completed | 343
Not completed — Adverse Event | 25
Not completed — Lack of Efficacy | 35
Not completed — Pregnancy | 5
Not completed — Lost to Follow-up | 82
Not completed — Subject Withdrew Consent | 92
Not completed — Protocol Violation | 60
Not completed — Other Miscellaneous Reasons | 43
Not completed — Missing | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Arm/Group | BOTOX®
Number analyzed (Participants) | 716
Age, Customized [Number; unit: participants]
  < 40 years | 270
  ≥ 40 years | 446
Gender [Count of Participants; unit: Participants]
  Female | 607
  Male | 109

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Frequency of Headache Days
Description: Mean change from Baseline in frequency (number) of headache days during the 28 day period ending with Week 108. A headache day was defined as a day (00:00 to 23:59) for which the participant reported a headache in the patient diary with 4 or more continuous hours of headache. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 108
Population: Analysis Population included all enrolled participants who had at least one efficacy assessment at baseline or a post-baseline visit.
Measure: Mean (Standard Deviation); unit: headache days
Arm/Group | BOTOX®
Number analyzed (Participants) | 715
headache days
  Baseline | 22.0 (4.82)
  Change from Baseline at Week 108 | -10.7 (6.44)

2. Secondary Outcome: Change From Baseline in the Frequency of Headache Days
Description: Mean change from Baseline in frequency (number) of headache days during the 28 day period ending with Week 60. A headache day was defined as a day (00:00 to 23:59) for which the participant reported a headache in the patient diary with 4 or more continuous hours of headache. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: headache days
Arm/Group | BOTOX®
Number analyzed (Participants) | 715
headache days
  Baseline | 22.0 (4.82)
  Change from Baseline at Week 60 | -9.2 (6.22)

3. Secondary Outcome: Change From Baseline in Headache Impact Test Questionnaire (HIT-6) Total Score
Description: The HIT-6 measures the impact of headache and treatment on the participant's functional health and well-being in 6 domains: pain; role functioning (ability to carry out usual activities); social functioning; energy or fatigue; cognition; and emotional distress assessed over the prior 4-week period. The total possible score ranges from 36 (no impact) to 78 (worst impact). A negative change from Baseline indicates an improvement, and a positive change from Baseline indicates a worsening.
Time Frame: Baseline, Week 60, Week 108
Population: Participants from the Analysis Population, all enrolled participants who had at least one efficacy assessment at baseline or a post-baseline visit, with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BOTOX®
Number analyzed (Participants) | 713
score on a scale
  Baseline | 64.7 (4.82)
  Change from Baseline at Week 60 | -6.8 (6.55)
  Change from Baseline at Week 108 | -7.1 (7.24)

ADVERSE EVENTS:
Time Frame: 108 Weeks
Description: Safety population included all participants who received at least one BOTOX® treatment injection.
Arm/Group | BOTOX®
Serious Adverse Events (participants affected / at risk) | 75/716
Other Adverse Events (participants affected / at risk) | 75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® (N=716)
Aortic valve incompetence (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Cushing's syndrome (Endocrine disorders) | 1
Cataract subcapsular (Eye disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Device intolerance (General disorders) | 1
Fatigue (General disorders) | 1
Non-cardiac chest pain (General disorders) | 3
Pyrexia (General disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Meningitis viral (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Ligament injury (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 2
Rib fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Obesity (Metabolism and nutrition disorders) | 1
Electrocardiogram abnormal (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Diabetic hyperosmolar coma (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 1
Intracranial hypotension (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 6
Paraesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 2
Suicidal ideation (Psychiatric disorders) | 5
Calculus ureteric (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Cholecystectomy (Surgical and medical procedures) | 1
Hysterectomy (Surgical and medical procedures) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | BOTOX®
Sinusitis (Infections and infestations) | 37/716
Neck pain (Musculoskeletal and connective tissue disorders) | 38/716

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that results publication or presentations be submitted for sponsor review no less than 90 days in advance, during which the sponsor can embargo such communications prior to public release. The embargo may be extended for up to 90 days for the sponsor to preserve its proprietary rights. PI will not publish study results prior to release of a multicenter manuscript including data from all study centers. The sponsor cannot require changes to the communication.